CLINICAL TRIAL: NCT02343172
Title: A Phase Ib/II, Open-label, Multicenter Study of Oral HDM201 in Combination With Oral LEE011 in Adult Patients With Liposarcoma
Brief Title: Study of Safety and Efficacy of HDM201 in Combination With LEE011 in Patients With Liposarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHDM201X2103C
Record Dates: First submitted 2015-01-05; First posted 2015-01-21 (Estimated); Last update posted 2020-12-09 (Actual); Status verified 2020-06

CONDITIONS: Liposarcoma
Keywords: Liposarcoma; MDM2 inhibition; cdk4 inhibition; HDM201; LEE011
MeSH Terms: conditions — Liposarcoma | interventions — siremadlin; ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HDM201+LEE011 (Experimental)
  Interventions: Drug: HDM201; Drug: LEE011

INTERVENTIONS:
Drug: HDM201
Drug: LEE011

SUMMARY:
To determine the MTD/RP2D of the HDM201 and LEE011 combination and evaluate whether the combination is safe and has beneficial effects in patients with liposarcoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically documented, locally advanced or metastatic WD/DD liposarcoma who have received at least one prior systemic therapy
* Patients with radiologic progression, defined by RECIST v.1.1, occurring while on/or within 6 months after last systemic treatment, prior to enrollment
* ECOG performance status of 0-1

Exclusion Criteria:

* Prior treatment with compounds with the same mode of action
* Patients with TP53 mutated tumors, if the molecular status is known
* Symptomatic central nervous system metastases
* Inadequate organ function
* Previous and concomitant therapy that precludes enrollment, as defined by protocol

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-03-13 (Actual); Primary Completion 2019-10-16 (Actual); Study Completion 2019-10-16 (Actual)

PRIMARY OUTCOMES:
Phase Ib: Incidence of Dose Limiting Toxicities (DLTs) during the first cycle of treatment. | 5 years
  DLTs in the first cycle of treatment.
Phase Ib: Exposure to HDM201 and LEE011 as measured by AUC 0-24h | 5 years
  as measured by AUC0-24h
Phase II: Progression free survival (PFS) | 5 years
  To assess the preliminary anti-tumor activity of HDM201 in combination with LEE011 in liposarcoma

SECONDARY OUTCOMES:
Phase Ib/II: Incidence and severity of AEs and SAEs | 5 years
  Run-in part to assess safety of HDM201 in combination with LEE011
Phase Ib/II: number of patients with dose interruptions and reduction | 5 years
  Run-in part To assess tolerability of HDM201 in combination with LEE011
Phase Ib/II: dose intensity | 5 years
  Run-in part To assess tolerability of HDM201 in combination with LEE011
Phase Ib/II: Pharmacokinetics (PK) parameters of HDM201 and LEE011: Cmax | 5 years
  Run-in part to evaluate PK parameters of HDM201 and LEE011
Phase Ib/II: Pharmacokinetics (PK) parameters of HDM201 and LEE011: Tmax | 5 years
  Run-in part to evaluate the PK parameters of HDM201 and LEE011
Phase Ib/II: Pharmacokinetics (PK) parameters of HDM201 and LEE011: AUClast | 5 years
  Run-in part to evaluate the PK parameters of HDM201 and LEE011
Phase Ib/II: Pharmacokinetics (PK) parameters of HDM201 and LEE011: AUCtau | 5 years
  Run-in part to evaluate the PK parameters of HDM201 and LEE011
Phase Ib/II: Changes from baseline of Pharmacodynamics (PD) markers in blood (GDF-15) | 5 years
  Run-in part measure of GDF-15 fold-change in protein levels (PD direct targets of p53) to assess PD changes from baseline in blood and a potential relationship with clinical outcome.
Phase Ib/II: Changes from baseline of Pharmacodynamics (PD) markers in tumor tissue (p21, MDM2) | 5 years
  Run-in part measure of p21 and MDM2 protein levels by IHC (H-Score) (p53 and CDK4 pathways) to assess changes from baseline of PD markers in tumor tissue and a potential relationship with clinical outcome.
Phase Ib/II: anti-tumor activity endpoint (BOR, PFS) | 5 years
  Run-in part to assess PD effect of HDM201 and LEE011 and a potential relationship with clinical outcome
Phase Ib: BOR, ORR and PFS as per RECIST v1.1, assessed by investigator | 5 years
  Run-in part to assess the preliminary anti-tumor activity of HDM201 in combination with LEE011 in liposarcoma
Phase II: BOR, ORR and PFS as per RECIST v1.1, assessed by investigator | 5 years
  Run-in part to further assess the anti-tumor activity of HDM201 in combination with LEE011 in liposarcoma

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- Novartis Investigative Site, Toronto, Ontario, Canada
- France (2):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Lyon
- Germany (2):
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Ulm
- Novartis Investigative Site, Singapore, Singapore
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: Results for CHDM201X2103C can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17708